CLINICAL TRIAL: NCT02470286
Title: A Phase1, Double-blind, Randomized, Placebo-control, Single Center, Single Dose Administration, Dose Escalation Study to Investigate the Pharmacokinetics, Safety and Tolerability of SA001 in Healthy Male Volunteers.
Brief Title: A Phase 1 Clinical Study to Investigate the Pharmacokinetics and Safety/Tolerability of SA001 in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samjin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SJSA001
Record Dates: First submitted 2015-06-01; First posted 2015-06-12 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- Cohort 1 (SA001 60mg or Placebo) (Experimental): 6 subjects receiving a single dose of 60mg SA001 and 2 subjects receiving placebo
  Interventions: Drug: SA001 60mg or Placebo
- Cohort 2 (SA001 120mg or Placebo) (Experimental): 6 subjects receiving a single dose of 120mg SA001 and 2 subjects receiving placebo
  Interventions: Drug: SA001 120mg or Placebo
- Cohort 3 (SA001 180mg or Placebo) (Experimental): 6 subjects receiving a single dose of 180mg SA001 and 2 subjects receiving placebo
  Interventions: Drug: SA001 180mg or Placebo
- Cohort 4 (SA001 240mg or Placebo) (Experimental): 6 subjects receiving a single dose of 240mg SA001 and 2 subjects receiving placebo
  Interventions: Drug: SA001 240mg or Placebo
- Cohort 5 (SA001 300mg or Placebo) (Experimental): 6 subjects receiving a single dose of 300mg SA001 and 2 subjects receiving placebo
  Interventions: Drug: SA001 300mg or Placebo

INTERVENTIONS:
Drug: SA001 60mg or Placebo — * Study Drug: SA001 60mg
  * Comparator: Placebo
  * Cohort 1 in the part 1 (Dose escalation study)
  Arms: Cohort 1 (SA001 60mg or Placebo)
Drug: SA001 120mg or Placebo — * Study Drug: SA001 120mg
  * Comparator: Placebo
  * Cohort 2 in the part 1 (Dose escalation study) and part 2 (Food effect study)
  Arms: Cohort 2 (SA001 120mg or Placebo)
Drug: SA001 180mg or Placebo — * Study Drug: SA001 180mg
  * Comparator: Placebo
  * Cohort 3 in the part 1 (Dose escalation study)
  Arms: Cohort 3 (SA001 180mg or Placebo)
Drug: SA001 240mg or Placebo — * Study Drug: SA001 240mg
  * Comparator: Placebo
  * Cohort 4 in the part 1 (Dose escalation study)
  Arms: Cohort 4 (SA001 240mg or Placebo)
Drug: SA001 300mg or Placebo — * Study Drug: SA001 300mg
  * Comparator: Placebo
  * Cohort 5 in the part 1(Dose escalation study) and part 2 (Food effect study)
  Arms: Cohort 5 (SA001 300mg or Placebo)

SUMMARY:
The purpose of this phase1 study is to investigate the pharmacokinetics, safety and tolerability of a single oral dose of SA001 and its active metabolite in healthy male volunteers.

DETAILED DESCRIPTION:
This study consists of Part 1 followed Part 2.

Part 1 (Dose escalation study, SA001 60mg~300mg dose group) The part 1 is a dose escalation study. The starting dose is SA001 60mg, and the maximum dose is 300mg. Each dose group is assigned to SA001 or Placebo in a ratio of 3:1. The pharmacokinetics, safety and tolerability of SA001 and its metabolite are investigated after a single oral administration on the fasting state.

Part 2 (Single dose and food effect study, SA001 120mg and 300mg dose group) The purpose of this part 2 is to evaluate the food effect of a high-fat diets(HFDs) on the single oral dose pharmacokinetics of SA001 and its metabolite.

ELIGIBILITY:
Inclusion Criteria:

1. 19 years to 45 years (Healthy male Korean)
2. Body weight of 55 to 90kg; and BMI of 18.0 to 27.0 kg/m^2
3. Subject who voluntarily agrees to participate in this study and has given a written informed consent, after fully understanding the detailed explanation of this study

Exclusion Criteria:

1. Subject with a disease history of any clinically significant condition as below.

   - Liver, Kidney, nervous system, immune system, respiratory system, endocrine system, tumor, cardiovascular disease or mental illness (mood disorder or obsessive-compulsive disorder etc.) etc.
2. Subject with a history of gastrointestinal disease (Crohn's disease, ulcer, acute or chronic pancreatitis, etc.) or gastrointestinal surgery (except simple appendicectomy or hernia surgery) that may affect the absorption of the study drug
3. Subject with a history of clinically significant hypersensitivity or hypersensitivity reactions to drugs (aspirin, antibiotics, etc.)
4. Serum ALT(SGPT)/AST(SGOT) >1.5×institutional upper limit normal (ULN)
5. eGFR< 90mL/min/1.73m^2
6. Systolic blood pressure <100 mmHg or >160 mmHg
7. Diastolic blood pressure <60 mmHg or >100 mmHg
8. Inadequate cardiac function confirmed by 12-lead ECG findings at screening as followings:

   * QTcF > 430msec (males)
   * PR interval > 200msec or < 110msec
   * QRS complex > 120msec
   * Evidence of 2nd- or 3rd-degree atrioventricular (AV) block
   * Pathologic Q waves (defined as Q-wave > 40msec or depth > 0.5mV)
   * Evidence of ventricular preexicitation, left bundle branch block (LBBB), right bundle branch block (RBBB, Incomplete RBBB)
9. Subject with risk factors for Torsade de pointes such as long QT syndrome, family history of sudden death, heart failure, hypokalemia, and arrhythmias
10. Subject with a history of drug abuse within 60 days prior to screening or who is positive for drugs of abuse in urine tests at screening
11. Subject who received any prescription drug or herbal medicine within 14 days prior to the first administration of the Investigational product
12. Subject who received any drugs such as

    * Prescription drug or herbal medicine within 14 days prior to the first administration of the investigational products
    * Over the counter (OTC) or vitamin within 7 days prior to the first administration of the investigational products
13. Subject who received other investigational products within 90 days prior to the first administration of the investigational products
14. Subject who continuously drink alcohol (more than 21 units/week, 1 unit = 10 g of pure alcohol) or cannot abstain from alcohol during the study period
15. Subject with history of smoking within 90 days prior to the first administration of the investigational products
16. Subject who cannot prohibit grapefruit/ caffeine-containing foods during the study period from 3 days before the first administration of the investigational products
17. Man of reproductive potential not willing to use contraceptive measures during the study period
18. Subject not eligible for study participation in the opinion of the investigator

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2015-09-18 (Actual); Study Completion 2015-09-30 (Actual)

PRIMARY OUTCOMES:
The incidence of treated related adverse event | Part1: Day-2(administration) to approximately Day 15 (Post study visit)
  Safety/Tolerability Assessment in the part 1

SECONDARY OUTCOMES:
Area under the curve (AUC) from time 0 to the time of the last quantifiable concentration (AUC0-tlast) of SA001 and its metabolite | Part1: predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, and 48 hours postdose, Part2: predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, and 48 hours postdose
Area under the curve (AUC) from time 0 extrapolated to infinity (AUC0-∞) of SA001 and its metabolite | Part1: predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, and 48 hours postdose, Part2: predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, and 48 hours postdose
Maximum observed plasma concentration (Cmax) of SA001 and its metabolite | Part1: predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, and 48 hours postdose, Part2: predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, and 48 hours postdose
Time to reach the maximum observed plasma concentration (tmax) of SA001 and its metabolite | Part1: predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, and 48 hours postdose, Part2: predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, and 48 hours postdose
t1/2 of SA001 and its metabolite | Part1: predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, and 48 hours postdose, Part2: predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, and 48 hours postdose
CL/F of SA001 and its metabolite | Part1: predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, and 48 hours postdose, Part2: predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, and 48 hours postdose
Vz/F of SA001 and its metabolite | Part1: predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, and 48 hours postdose, Part2: predose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 32, and 48 hours postdose
CLR of SA001 and its metabolite | Part1: predose and 0 ~ 4, 4 ~ 8, 8 ~ 12, 12 ~ 24, 24 ~ 32 and 32 ~ 48 hours postdose, Part2: predose and 0 ~ 4, 4 ~ 8, 8 ~ 12, 12 ~ 24, 24 ~ 32 and 32 ~ 48 hours postdose
  CLR = Ae / AUCinf (Ae: total amount excreted in the urine)
Fraction recovered unchanged in urine (FR) of SA001 and its metabolite | Part1: predose and 0 ~ 4, 4 ~ 8, 8 ~ 12, 12 ~ 24, 24 ~ 32 and 32 ~ 48 hours postdose, Part2: predose and 0 ~ 4, 4 ~ 8, 8 ~ 12, 12 ~ 24, 24 ~ 32 and 32 ~ 48 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-sang Yu, M.D., Ph.D., M.B.A, Principal Investigator — Seoul National University College of Medicine / Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea